CLINICAL TRIAL: NCT01126931
Title: Pilot Trial With Wormwood to Improve Appetite in Cancer, Autoimmune Diseases, Depression and Old Age
Brief Title: Wormwood in Chronic Progressive Disorders With Reduced Appetite
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Freiburg (Other)
Responsible Party: Simone Krebs MD, Medical Faculty, University of Saarland, Homburg, Germany
Other Study IDs: Appetite and Weight Loss
Record Dates: First submitted 2010-05-17; First posted 2010-05-20 (Estimated); Last update posted 2010-05-20 (Estimated); Status verified 2008-02

CONDITIONS: Cancer
Keywords: Crohn disease; Involuntary weight loss in cancer; IgA nephropathy; Depression with reduced appetite
MeSH Terms: conditions — Neoplasms; Crohn Disease; Glomerulonephritis, IGA

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Wormwood is approved herbal medicine for the treatment of reduced appetite in Germany (Registration No.: 1339.99.99). Reduced appetite is observed in many chronic health disorders such as old age, immune disorders and cancer.

Trial aims at observing beneficial effects of wormwood supplementation in various chronic disorders associated with reduced appetite

DETAILED DESCRIPTION:
Supplementation with wormwood in chronic disorders associated with reduced appetite.

Examples:

1. Cancer
2. Autoimmune diseases such as Crohns disease and IgA Nephropathy
3. Old age
4. Chronic stress and depression

ELIGIBILITY:
Inclusion Criteria:

* Appetite and weight loss
* Chronic progressive disease

Exclusion Criteria:

* Life expectancy less than 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with reduced appetite and reduced quality of life as a result of chronic progressive disorders such as cancer, autoimmune diseases (Crohn, IgA-Nephropathy), old age and depression
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2006-02; Primary Completion 2012-08 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Improvement in appetite | 6-12 months

SECONDARY OUTCOMES:
Improvement in quality of life | 12-24 months

CONTACTS AND LOCATIONS:
Overall Officials: Simone S Krebs, MD, PhD, Principal Investigator — University of Freiburg, Nuclear Medicine, Germany
Locations (1):
- University of Freiburg, Medical Faculty, Freiburg im Breisgau, Baden, Germany

REFERENCES:
- [Background] Omer B, Krebs S, Omer H, Noor TO. Steroid-sparing effect of wormwood (Artemisia absinthium) in Crohn's disease: a double-blind placebo-controlled study. Phytomedicine. 2007 Feb;14(2-3):87-95. doi: 10.1016/j.phymed.2007.01.001. Epub 2007 Jan 19. PMID 17240130
- [Background] Krebs S, Omer TN, Omer B. Wormwood (Artemisia absinthium) suppresses tumour necrosis factor alpha and accelerates healing in patients with Crohn's disease - A controlled clinical trial. Phytomedicine. 2010 Apr;17(5):305-9. doi: 10.1016/j.phymed.2009.10.013. Epub 2009 Dec 3. PMID 19962291
- [Derived] Krebs S, Omer B, Omer TN, Fliser D. Wormwood (Artemisia absinthium) for poorly responsive early-stage IgA nephropathy: a pilot uncontrolled trial. Am J Kidney Dis. 2010 Dec;56(6):1095-9. doi: 10.1053/j.ajkd.2010.06.025. Epub 2010 Sep 16. PMID 20843592